CLINICAL TRIAL: NCT04372810
Title: Acute Effect of Manual Therapy on Tibiotarsal Joint Mobility of Lower Limbs in Diabetic Individuals
Brief Title: Effect of Manual Therapy on Tibiotarsal Joint Mobility in Diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 63957816.7.0000.5440
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Complications
Keywords: Physiotherapy; Diabetes Melittus; Manual Therapy; Ankle Joint
MeSH Terms: conditions — Diabetes Complications | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The volunteers were randomized by means of sealed matte envelopes in the following groups: sham group (GS), evaluated on day 1 and day 7, and received preventive diabetes guidance at the end of the experiment (follow-up) and intervention group (GI), assessed on day 1, then underwent manual manipulation intervention and were reevaluated post-intervention. They were again evaluated on the 7th post-treatment day and received preventive guidance at the end of the experiment (follow-up).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group, assessed on day 1, then underwent manual manipulation intervention and were reevaluated post-intervention and again evaluated on the 7th post-treatment day and received preventive guidance at the end of the experiment (follow-up).
  Interventions: Procedure: High Velocity Low Amplitude manipulation (HVLA); Procedure: Care assessment and guidance
- Sham Group (Sham Comparator): Sham group, evaluated on day 1 and day 7, and received preventive diabetes guidance at the end of the experiment (follow-up).
  Interventions: Procedure: Care assessment and guidance

INTERVENTIONS:
Procedure: High Velocity Low Amplitude manipulation (HVLA) — The thrust manipulation technique was used, which consists of high speed and small amplitude manipulation. The therapeutic intervention was performed through decompressive maneuvers for the tibiotarsal joints. The choice of the place of application of the manipulation technique was delimited by the identification of the area or areas with compressive compartmental impairment and joint restriction. The use of the method depended directly on the identification of one or more regions of joint restraint.
  Arms: Intervention Group
Procedure: Care assessment and guidance — Evaluation and care guidelines on glycemic control and diabetic foot care.

SUMMARY:
The study aimed to evaluate the acute effect of manual therapy on ankle joint mobility in diabetic patients. Forty volunteers, with a mean age of 59.35±7.85, with type 2 DM and neurological symptoms of Diabetic Distal Polyneuropathy according to a Diabetic Polyneuropathy Diagnostic Scale (EDPNDD) protocol with the amplitude were performed. Were divided into two groups: Sham group (GS), and intervention group (GI), which underwent manual manipulation intervention and seven-day follow-up. Joint range of motion analysis was performed using digital goniometry and static discharge of weights assessed by computerized baropodometry with open and closed eyes, and the Shapiro-Wilk normality test evaluated data distribution and relative, Tukey post hoc set ANOVA tests were used for non-normal variables. The Kruskal- Wallis test followed by Dunn's post-hoc test. SAS statistical software was used and the significance level of 5%. Results: The results showed an increased joint range of motion, plantar flexion, and dorsiflexion, between the moments and moments after manipulation and follow-up. It was still possible to make a significant difference between GI when it was with GS at poster and follow-up. No intragroup analysis was performed by GS, for analysis over time. Regarding intragroup comparisons over time (pre, post-intervention, and follow-up), a significant difference was made for Front and back displacement amplitude (PAD) with open eyes of the GI, with an increase after intervention and reduction without follow up. Conclusion: Based on the results obtained, the work performed with manual therapy increased the ankle joint amplitude in diabetic individuals.

DETAILED DESCRIPTION:
Diabetes Melittus (DM) is a disease of great incidence, and one of the main public health problems worldwide, having as complications the deficit in the functional performance of the lower limbs, which can interfere in the maintenance of the balance, besides being a Strong predictor of functional limitations. Individuals affected by diabetes are predisposed to reduce the mobility of the tibial-tarsal joint. Manual therapy is often used for the purpose of improving range of motion. The objective of this study is to evaluate the acute effect of manual therapy on ankle joint mobility in diabetic patients. 40 volunteers, aged 59,35±7,85 years, DM type 2 and tibial-tarsal joint amplitude limitation, of both genders were recruited, divided into two groups: group 1 (Sham: submitted to evaluations and follow up of seven days), and group 2 (intervention: submitted to the evaluations, manipulative manual intervention, with follow up of seven days). The analysis of joint range of motion was acessed by digital goniometry and the static discharge of weight was evaluated by baropodometry computed with open and closed eyes. After tabulation of variables, the Shapiro-Wilk normality test was applied to analyze the distribution. Before a normal and related distribution, ANOVA followed by Tukey post-hoc tests were used. For the variables that presented a non-normal distribution, the Kruskal-Wallis test was used, followed by the Dunn post-hoc test. For the variables that presented a non-normal distribution, the Kruskal-Wallis test was used, followed by the Dunn post-hoc test. The SAS software was used and a significance level of 5% was considered. The results showed an increase in joint range of motion, in the right and left dorsiflexions of the GI between the initial moment and the post-manipulation moments, as well as after seven days of the follow-up. There was also a significant difference between GI when compared to GS in the post and follow-up moments. Regarding the clinical effect of the intervention over time, the intragroup analysis showed that in GS there was no difference between the amplitude of movement registers comparing the pre-intervention moment with the subsequent records (post and follow-up), even for plantar and dorsiflexion flexion movements on both sides. In relation to static plantar weight discharge, there was a change in recorded values for the peak of total foot pressure, on the right and left sides of the GI, between the moments after the immediate intervention and in the measurement 7 days after the manipulative intervention (follow -up), for registration with open eyes. Regarding intra-group comparisons over time (pre, post-intervention and follow-up), a significant difference was observed for the condition amplitude of anteroposterior displacement (DAP) with open eyes of the GI, observing an increase after intervention and reduction in the follow-up. In view of the obtained results, it can be inferred that the acute intervention with manual therapy produces an increase in the joint amplitude of the ankle of diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes aged between 35 and 70 years, and with more than 5 years of Diagnosis of Diabetes Mellitus.

Exclusion Criteria:

Patients with skin lesions or lower limb fractures in the last six months, plantar malformations, severe postural changes and real difference in the length of the lower limbs.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Tibiotarsal joint range of motion | 2 minutes
  degrees

SECONDARY OUTCOMES:
Static balance | 6 minute
  cm

CONTACTS AND LOCATIONS:
Overall Officials: Elaine CO Guirro, PhD, Study Director — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Medical School of Ribeirão Preto, Ribeirão Preto, São Paulo
  - University of São Paulo, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No
after the end of Research

REFERENCES:
- [Result] Marron-Gomez D, Rodriguez-Fernandez AL, Martin-Urrialde JA. The effect of two mobilization techniques on dorsiflexion in people with chronic ankle instability. Phys Ther Sport. 2015 Feb;16(1):10-5. doi: 10.1016/j.ptsp.2014.02.001. Epub 2014 Feb 14. PMID 24679362